CLINICAL TRIAL: NCT04065789
Title: Safety, Tolerability, and Efficacy of Once Weekly Carfilzomib in Combination With Daratumumab, Lenalidomide and Dexamethasone, in Transplant-ineligible Multiple Myeloma Patients Non-responsive to a Bortezomib Based Induction
Brief Title: Carfilzomib in Combination With Daratumumab, Lenalidomide and Dexamethasone in Transplant-ineligible NDMM Patients
Acronym: KyDaR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0101-17-TLV; MOH_2018-01-18_001958 (Other: Israel MOH#)
Record Dates: First submitted 2019-07-31; First posted 2019-08-22 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Myeloma Multiple; Myeloma, Plasma-Cell; Myeloma-Multiple; Plasma Cell Myeloma
Keywords: multiple myeloma (MM); Myeloma; NDMM; RRMM
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — carfilzomib; daratumumab; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Carfilzomib,Daratumumab,revlimid and dexamethasone (Experimental): Carfilzomib, Daratumumab, Lenalidomide, Dexamethasone
  Interventions: Drug: Carfilzomib; Drug: Daratumumab; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib — Carfilzomib on Days 1, 8, 15, of cycle numbers 1-9 and Days 1 and 15 only of cycle numbers 10-18, at a dose of 20 mg/m2 on day 1 of cycle 1; at dose of 56 mg/m2 on all subsequent once weekly dosing days. The quadruple regimen treatment will be administered for 18 cycles.
  Other Names: Kyprolis
Drug: Daratumumab — Daratumumab : 16 mg/Kg weekly for 8 weeks, then every 2 weeks for 16 weeks, and then every 4 weeks thereafter. The quadruple regimen treatment will be administered for 18 cycles.
  Other Names: Darzalex
Drug: Lenalidomide — Lenalidomide (25 mg), administered on days 1-21 of 28-day cycle.In frail patients, Lenalidomide dose will be reduced according to 15 mg . The quadruple regimen treatment will be administered for 18 cycles.
  Other Names: Revlimid
Drug: Dexamethasone — Patients will be treated with IV or oral dexamethasone (20 mg for fit and INT-FIT, 10 mg for frail), administered on Days 1-2, 8-9, 15-16, and 22-23 of each 28-day cycle for cycles 1-2 followed by weekly 20 mg dexamethasone on subsequent cycles; In frail patients, dexamethasone will be reduced to 10 mg . The quadruple regimen treatment will be administered for 18 cycles.

SUMMARY:
Patients with newly diagnosed multiple myeloma (NDMM) who failed to achieve at least a minimal response (MR) after 2 cycles or a partial response (PR), after 4 cycles of a bortezomib-containing therapy, or progress on therapy during first 4 cycles (response defined by international Myeloma Working Group [IMWG] criteria), will be treated with a quadruple regimen comprised of: Daratumumab 16 mg/Kg weekly during cycles 1-2, q14 days during cycles 3-6, thereafter monthly (1st dose cycle 1 may be split over 2 days); Once-weekly intravenous (IV) administration of Carfilzomib on days 1, 8, 15, of cycle numbers 1-9 and Days 1 and 15 only of cycle numbers 10-18, at a dose of 20 mg/m2 on day 1 of cycle 1; at dose of 56 mg/m2 on all subsequent once weekly dosing days, alongside concomitant treatment with twice-weekly IV or oral dexamethasone 20mg administered on Days 1-2, 8-9, 15-16, and 22-23 of a 28-day cycle, for cycles 1-2 followed by weekly 20 mg dexamethasone on subsequent cycles; and oral Lenalidomide 25 mg, administered on days 1-21 of a 28-day cycle. On treatment days that require both Carfilzomib and Daratumumab infusions, Carfilzomib will be administrated prior to Daratumumab administration. All patients will undergo frailty assessment based on IMWG recommendations, and will be classified as fit, intermediate-fit and frail. Frail patients will receive Lenalidomide dose adjustment to 15 mg (throughout the study, from cycle 1 and on), and dexamethasone at 10 mg x 2/week cycles 1-2 followed by 10 mg/week for subsequent cycles. The quadruple regimen will be administered for 18 cycles, followed by long-term follow-up in which patients will receive standard of care treatment with Lenalidomide/dexamethasone (Rd) treatment, unless disease progression, the physician decides otherwise, the patient suffers from unacceptable toxicity, withdraws consent, or dies (whichever occurs first).

DETAILED DESCRIPTION:
Patients with newly diagnosed multiple myeloma (NDMM) who failed to achieve at least a minimal response (MR) after 2 cycles or a partial response (PR), after 4 cycles of a bortezomib-containing therapy, or progress on therapy during first 4 cycles (response defined by international Myeloma Working Group [IMWG] criteria), will be treated with a quadruple regimen comprised of: Daratumumab 16 mg/Kg weekly during cycles 1-2, q14 days during cycles 3-6, thereafter monthly (1st dose cycle 1 may be split over 2 days); Once-weekly intravenous (IV) administration of Carfilzomib on days 1, 8, 15, of cycle numbers 1-9 and Days 1 and 15 only of cycle numbers 10-18, at a dose of 20 mg/m2 on day 1 of cycle 1; at dose of 56 mg/m2 on all subsequent once weekly dosing days, alongside concomitant treatment with twice-weekly IV or oral dexamethasone 20mg administered on Days 1-2, 8-9, 15-16, and 22-23 of a 28-day cycle, for cycles 1-2 followed by weekly 20 mg dexamethasone on subsequent cycles; and oral Lenalidomide 25 mg, administered on days 1-21 of a 28-day cycle. On treatment days that require both Carfilzomib and Daratumumab infusions, Carfilzomib will be administrated prior to Daratumumab administration. All patients will undergo frailty assessment based on IMWG recommendations, and will be classified as fit, intermediate-fit and frail. Frail patients will receive Lenalidomide dose adjustment to 15 mg (throughout the study, from cycle 1 and on), and dexamethasone at 10 mg x 2/week cycles 1-2 followed by 10 mg/week for subsequent cycles. The quadruple regimen will be administered for 18 cycles, followed by long-term follow-up in which patients will receive standard of care treatment with Lenalidomide/dexamethasone (Rd) treatment, unless disease progression, the physician decides otherwise, the patient suffers from unacceptable toxicity, withdraws consent, or dies (whichever occurs first). All patients will be required to receive either thromboprophylaxis or anticoagulation therapy in parallel. Patients will receive prophylaxis to herpes zoster and pneumocystis infection according to institutional guidelines, as well as proton pump inhibitors on dexamethasone treatment days only, according to institutional guidelines.

Patients will be assessed for response, to be determined by multiple myeloma (MM) biomarker profiling, on day 1 of cycle 2 and then every 56 ±4 days thereafter, irrespective of treatment delays or the timing of treatment cycles. Disease status will be followed until confirmed progressive disease (PD).

Long-term follow-up for disease status (only in cases where patients discontinued treatment prior to PD or patients completing all 18 cycles without signs of PD) and for survival (after reaching PD) will continue after treatment discontinuation until the patient has withdrawn consent for further participation, is lost to follow-up, has died, or the sponsor makes a decision to terminate the study. For patients who discontinued treatment before completing 18 cycles , without PD occurred, disease response assessments shall be performed every 56 days (±4 days), according to the original scheduled days of assessment, until disease progression. Patients completing all 18 cycles without signs of PD will be followed-up for disease response every 84±7 days. Follow-up for survival will be performed approximately every 3 months, or as needed, for all surviving patients until study closure. For any patient who is lost to follow-up, the study site will attempt to ascertain survival information via public database search.

The control group in this study (Historical Control) will consist of 144 consecutive patients from a subset of participating centers and will include transplant ineligible NDMM diagnosed between 2011 to 2017 with failure to respond to a bortezomib based induction (as defined in the prospective trial). Control group patients must meet the protocol inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with multiple myeloma and started induction therapy within 6 months prior to study entry
2. Received bortezomib-based induction therapy, with corticosteroids, with or without alkylators
3. Determined by investigator to be transplant-ineligible
4. Failed to achieve a minimal response (MR) after 2 cycles or a partial response (PR), after 4 cycles of a bortezomib-containing therapy, or progress on therapy during first 4 cycles (response defined by international Myeloma Working Group [IMWG] criteria)
5. Measurable disease at time of enrolment including:

   * Serum M-protein ≥ 0.5 g/dL, or
   * Urine M-protein ≥ 200 mg/24 hour, or
   * Serum free light chain (SFLC) ≥ 100 mg/L (involved light chain) and an abnormal serum kappa/lambda ratio, or
   * In patients with immunoglobulin A (IgA) type MM, whose disease can only be reliably measured by serum quantitative immunoglobulin (qIgA), qIgA ≥ 750 mg/dL (0.75 g/dL)
6. Male/female, ≥ 18 years of age
7. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0-2
8. Adequate hepatic function within 28 days prior to treatment initiation, with bilirubin < 1.5 times the upper limit of normal (ULN), and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 times the ULN
9. Left ventricular ejection fraction ≥ 40%
10. Absolute neutrophil count (ANC) ≥ 1500/mm3 within 28 days prior to enrollment, and reconfirmed within 7 days prior to first dose. Screening ANC should be independent of growth factor support for ≥ 1 week.
11. Hemoglobin ≥ 8.0 g/dL within 28 days prior to treatment initiation, and reconfirmed within 7 days prior to first dose. Use of erythropoietic stimulating factors and red blood cell (RBC) transfusions per institutional guidelines is allowed, however most recent RBC transfusion may not have been done within 7 days of obtaining Screening hemoglobin.
12. Platelet count ≥ 50,000/mm3 (≥ 30,000/mm3 if myeloma involvement in the bone marrow is > 50%) within 28 days prior of treatment initiation, and reconfirmed within 7 days prior to first dose. Patients should not have received platelet transfusions for at least 1 week prior to obtaining the Screening platelet count.
13. Calculated or measured creatinine clearance (CrCL) of ≥ 30 mL/min within 28 days prior to treatment initiation. Calculation should be based on standard formula such as the Cockcroft and Gault: [(140 - Age) x Mass (kg) / (72 x Creatinine mg/dL)]; multiply result by 0.85 if female.
14. Written informed consent in accordance with local regulations
15. Females of childbearing potential (FCBP) must have a negative serum pregnancy test within 21 days prior to treatment initiation and agree to use an effective method of contraception throughout the treatment period and for 3 months following last dose. Female of childbearing potential is defined as a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy or 2) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
16. Male patients must use an effective barrier method of contraception during the treatment period and for 3 months following the last dose, if sexually active with a FCBP -

Exclusion Criteria:

1. Prior therapy with any immunomodulatory drug (IMiD) or with Carfilzomib
2. Any unresolved Grade 2 or higher toxicity from bortezomib based induction treatment
3. Multiple myeloma of immunoglobulin M (IgM) subtype
4. POEMS (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes) syndrome
5. Plasma cell leukemia or circulating plasma cells ≥ 2 × 10e9/L
6. Waldenström macroglobulinemia
7. Patients with known amyloidosis
8. Focal radiation therapy within 7 days prior to treatment initiation; radiation therapy to an extended field, involving a significant volume of bone marrow, within 21 days prior to enrollment (i.e., prior radiation must have been to less than 30% of the bone marrow)
9. Major surgery (excluding kyphoplasty) within 28 days prior to treatment initiation
10. Active congestive heart failure (New York Heart Association [NYHA] Class III to IV), symptomatic ischemia, or conduction abnormalities uncontrolled by conventional intervention; myocardial infarction within 4 months prior to treatment initiation
11. Acute active infection requiring systemic antibiotics, antiviral (except antiviral therapy directed at hepatitis B) or antifungal agents within 14 days prior to treatment initiation
12. Known human immunodeficiency virus (HIV) seropositive, hepatitis C infection, and/or hepatitis B (except for patients with hepatitis B surface antigen [SAg] and core antibody receiving and responding to antiviral therapy directed at hepatitis B; these patients are allowed).
13. Patients with known cirrhosis
14. Second malignancy within the past 3 years except:

    A. Adequately treated basal cell or squamous cell skin cancer B. Carcinoma in situ of the cervix C. Prostate cancer Gleason score ≤ 6 with stable prostate-specific antigen (PSA) over 12 months D. Breast carcinoma in situ with full surgical resection E. Treated medullary or papillary thyroid cancer
15. Patients with myelodysplastic syndrome
16. Female patients who are pregnant or lactating
17. Known history of allergy to Captisol (a cyclodextrin derivative used to solubilize Carfilzomib)
18. Patients with hypersensitivity to Carfilzomib,
19. Contraindication to any of the required concomitant drugs or supportive treatments, including hypersensitivity to antiviral drugs, or intolerance to hydration due to pre-existing pulmonary or cardiac impairment
20. Patients with pleural effusions requiring thoracentesis or ascites requiring paracentesis within 14 days prior to treatment initiation
21. Subject has either one of the following:

    1. Known chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) <50% of predicted normal. Note that FEV1 testing is required for subjects suspected of having COPD and subjects must be excluded if FEV1 is <50% of predicted normal.
    2. Known moderate or severe persistent asthma, within the past 2 years, uncontrolled asthma of any classification. Note that subjects who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed to participate in the study.
22. Patients who discontinued bortezomib due to bortezomib related adverse events.
23. Any other clinically significant medical disease or psychiatric condition that, in the investigator's opinion, may interfere with protocol adherence or a patient's ability to give informed consent
24. Any prior treatment with investigational anti-MM drugs -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2021-11-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who experience any AE incidence, grade > 2 drug-elicited toxicities, peripheral neuropathy events (Grade 2 or higher). | from screening through month 20
  Determined by adverse events, vital signs and clinical laboratory parameters in relation to study intervention.

SECONDARY OUTCOMES:
PFS | From treatment initiation to the earlier of disease progression or death due to any cause. Up to 2 years from last patient enrollment
  Progression Free Survival (PFS)
OS | From treatment initiation to date of death (whatever the cause). Up to 2 years from last patient enrollment
  Overall Survival (OS)
Overall response rate (ORR) | From Screening and up to 2 years from last patient enrollment
  The fraction of patients who experience a partial response (PR), very good partial response (VGPR), complete response (CR), or stringent complete response (sCR) per IMWG 2016 criteria.
Duration of response (DOR) | From initiation of treatment and up to 2 years from last patient enrollment
  Time of first evidence of PR or better to confirmation of PD or death due to any cause
Time to progression (TTP) | From initiation of treatment and up to 2 years from last patient enrollment
  From initiation of treatment to documented PD
Clinical benefit response (CBR) rate | From initiation of treatment and up to 2 years from last patient enrollment
  Defined as ORR or minimal response (MR)
Disease control rate (DCR), | From initiation of treatment and up to 2 years from last patient enrollment
  Defined as ORR or minimal response (MR) or stable disease (SD) lasting at least 8 weeks.
Changes in Global Health Status and Quality of Life | From Screening and up to 2 years from last patient enrollment
  The European Organization for Research and Treatment of Cancer [EORTC] Quality of Life Questionnaire Module QLQ-MY20 will be used to evaluate Global Health Status/QoL. Questionnaire Module QLQ-MY20 include 20 questions (items). Score scale is starting from minimum of 1 and up to a maximum of 4. Higher values represent a worse outcome.It is the complementary module of the QLQ-C30 which is specific for Multiple Myeloma patients.
Changes in Global Health Status and Quality of Life | From Screening and up to 2 years from last patient enrollment
  The European Organization for Research and Treatment of Cancer [EORTC] Quality of Life Questionnaire Module QLQ-C30 will be used to evaluate Global Health Status/QoL. Questionnaire Module QLQ-C30 include 30 questions score scale is starting from minimum of 1 and up to a maximum of 7. In most items (1-28) Higher values represent a worse outcome.The exceptions are the items contributing to the global health status / QoL - 2 items (29-30) In which Higher values represent a better outcome .
  It incorporates five functional scales (physical, role, cognitive, emotional, and social), three symptom scales (fatigue, pain, and nausea and vomiting), a global health status / QoL scale, and a number of single items assessing additional symptoms commonly reported by cancer patients (dyspnoea, loss of appetite, insomnia, constipation and diarrhoea) and perceived financial impact of the disease.
Changes in Frailty Status | From Screening and up to 4 month from last patient enrollment
  Frailty assessment, for this study will be based only on 4 components : age, the Charlson Comorbidity Scoring System, the Katz Index of Independence in Activities of Daily Living and the Lawton Instrumental Activities of Daily Living Scale.
  All above 4 components are summed up and combined into one MM Frailty score - The score system (range 0-5, higher values represent a worse outcome), identifies 3 groups of patients:
  fit (score=0) intermediate-fitness (score=1) frail (score≥2)

OTHER OUTCOMES:
exploratory genomic profiling | From Screening and up to 2 years from last patient enrollment
  mutational transcriptional and post translational changes associated with drug sensitivity and resistance, clonal evolution

CONTACTS AND LOCATIONS:
Overall Officials: Yael Cohen, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (14):
- Israel (14):
  - Haemek Medical Center, Afula
  - Barzilai Medical Center, Ashkelon
  - Soroka Medical Center, Beersheba
  - Bnai-Zion Medical Center, Haifa
  - Carmel Medical center, Haifa
  - Rambam medical Center, Haifa
  - Hadassah Ein-Karem Medical Center, Jerusalem
  - Shaare Zedek medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Kaplan Medical center, Rehovot
  - Ziv Medical Center, Safed
  - Hematology Department Sourasky Medical Center, Tel Aviv
  - Assuta Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cohen YC, Zada M, Wang SY, Bornstein C, David E, Moshe A, Li B, Shlomi-Loubaton S, Gatt ME, Gur C, Lavi N, Ganzel C, Luttwak E, Chubar E, Rouvio O, Vaxman I, Pasvolsky O, Ballan M, Tadmor T, Nemets A, Jarchowcky-Dolberg O, Shvetz O, Laiba M, Shpilberg O, Dally N, Avivi I, Weiner A, Amit I. Identification of resistance pathways and therapeutic targets in relapsed multiple myeloma patients through single-cell sequencing. Nat Med. 2021 Mar;27(3):491-503. doi: 10.1038/s41591-021-01232-w. Epub 2021 Feb 22. PMID 33619369